CLINICAL TRIAL: NCT04176354
Title: Real-world Treatment Patterns and Effectiveness of Palbociclib in Combination With an Aromatase Inhibitor as Initial Endocrine Based Therapy in Metastatic/Advanced Breast Cancer
Brief Title: Real-world Treatment Patterns and Effectiveness of Palbociclib and AI Therapy
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481122
Record Dates: First submitted 2019-10-24; First posted 2019-11-25 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Palbociclib; Real-world data; Retrospective study; Effectiveness
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Palbociclib + an aromatase inhibitor: Adult metastatic breast cancer patients who initiated Palbociclib + an aromatase inhibitor as first line therapy between Feb 3, 2015 to 3 months prior to date of data cutoff in the Flatiron Health Analytic Database.
  Interventions: Drug: Palbociclib + an aromatase inhibitor
- Palbociclib + Letrozole: Adult metastatic breast cancer patients who initiated Palbociclib +Letrozole as first line therapy between Feb 3, 2015 to 3 months prior to date of data cutoff in the Flatiron Health Analytic Database.
  Interventions: Drug: Palbociclib + Letrozole
- Letrozole: Adult metastatic breast cancer patients who initiated Letrozole as first line therapy between Feb 3, 2015 to 3 months prior to date of data cutoff in the Flatiron Health Analytic Database.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib + an aromatase inhibitor — Palbociclib + an aromatase inhibitor therapy
  Groups: Palbociclib + an aromatase inhibitor
Drug: Palbociclib + Letrozole — Palbociclib + Letrozole therapy
  Groups: Palbociclib + Letrozole
Drug: Letrozole — Letrozole monotherapy
  Groups: Letrozole

SUMMARY:
A retrospective observational analysis of de-identified Flatiron Health Analytic Database to describe patient characteristics, treatment patterns and effectiveness of Palbociclib + AI as first-line therapy in HR+/HER2- metastatic breast cancer (MBC) in the US clinical practices.

DETAILED DESCRIPTION:
Utilizing de-identified data derived from the Flatiron Health Analytic Database, the retrospective observational study is to describe patient characteristics, treatment patterns and effectiveness of Palbociclib + AI as first-line therapy in HR+/HER2-MBC in the US real-world clinical practice setting. Patients will be evaluated retrospectively from index therapy date to death, or last visit in the database, whichever comes first. Descriptive and multivariate statistical analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex
2. At least 18 years old at MBC diagnosis
3. Diagnosis of MBC at any point in patient history

   1. ICD-9 (174.x, 175.x) or ICD-10 (C50.xx) diagnosis of BC
   2. Confirmation of metastatic disease
   3. At least 2 document clinical visits
   4. Evidence of stage IV or recurrent MBC with a metastatic diagnosis date on or after 2011, as confirmed by unstructured clinical documents
4. HR+/HER2-

   1. HR+: ER+ or PR+ test before or up to 60 days after MBC diagnosis
   2. HER2-: any HER2 negative test and the absence of a positive test (IHC positive 3+, FISH positive/amplified, Positive NOS) before or up to 60 days after MBC diagnosis
5. Palbociclib + AI or letrozole as first-line therapy for MBC during the period from February/2015 through August /31/2018 (or 3 months prior to study cut-off date) to allow for a possible minimum follow-up time of 90 days until the study cutoff date. AI was administered within (±) 28 days of Palbociclib index date.

Exclusion Criteria:

1. Evidence of prior treatment with other CDK4/6I (Ribociclib or Abemaciclib), AI (Letrozole, Exemestane, and Anastrazole), Tamoxifen, Raloxifene, Toremifene, or Fulvestrant for MBC
2. First structured activity greater than 90 days after MBC diagnostic date
3. Treatment with a CDK4/6 inhibitor as part of a clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HR+/HER2- MBC female adult patients treated with Palbociclib + AI or Letrozole alone between February2015 and end of 2018 or data cut-off date
Sampling Method: Non-Probability Sample
Enrollment: 813 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Brufsky A, Liu X, Li B, McRoy L, Layman RM. Real-World Effectiveness of Palbociclib Plus Letrozole vs Letrozole Alone for Metastatic Breast Cancer With Lung or Liver Metastases: Flatiron Database Analysis. Front Oncol. 2022 Jul 4;12:865292. doi: 10.3389/fonc.2022.865292. eCollection 2022. PMID 35860587
- [Derived] Patt D, Liu X, Li B, McRoy L, Layman RM, Brufsky A. Real-World Treatment Patterns and Outcomes of Palbociclib Plus an Aromatase Inhibitor for Metastatic Breast Cancer: Flatiron Database Analysis. Clin Breast Cancer. 2022 Aug;22(6):601-610. doi: 10.1016/j.clbc.2022.05.002. Epub 2022 May 5. PMID 35643624
- [Derived] Brufsky A, Liu X, Li B, McRoy L, Layman RM. Real-World Tumor Response of Palbociclib Plus Letrozole Versus Letrozole for Metastatic Breast Cancer in US Clinical Practice. Target Oncol. 2021 Sep;16(5):601-611. doi: 10.1007/s11523-021-00826-1. Epub 2021 Aug 2. PMID 34338965
- [Derived] DeMichele A, Cristofanilli M, Brufsky A, Liu X, Mardekian J, McRoy L, Layman RM, Emir B, Torres MA, Rugo HS, Finn RS. Comparative effectiveness of first-line palbociclib plus letrozole versus letrozole alone for HR+/HER2- metastatic breast cancer in US real-world clinical practice. Breast Cancer Res. 2021 Mar 24;23(1):37. doi: 10.1186/s13058-021-01409-8. PMID 33761995
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481122

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with hormone receptor positive(HR+)/human epidermal growth factor receptor 2negative (HER2-)metastatic breast cancer(MBC),who received palbociclib in combination with aromatase inhibitor(AI)[letrozole,anastrozole or exemestane]during 03-February-2015 to 31-August-2018(approximately 3.6years)were observed retrospectively.
Pre-assignment Details: Data of participants was retrieved from Flatiron Health Analytic database. Available data was evaluated in 9 months of retrospective observational study.
Groups:
- Palbociclib + AI: Participants who received palbociclib in combination with AI under standard real world clinical practice for HR+/HER2- MBC during the period 03-February-2015 to 31-August-2018 were included in this retrospective observational study. Available data were evaluated in 9 months of this retrospective, observational study.
Period: Overall Study
Arm/Group | Palbociclib + AI
Started | 813
Completed | 813
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Arm/Group | Palbociclib + AI
Number analyzed (Participants) | 813
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 813
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 555
  Black | 63
  Asian | 18
  Hispanic or Latino | 23
  Other/Unknown | 154

OUTCOME MEASURES:

1. Primary Outcome: Real-World Progression Free Survival (rwPFS): Using Kaplan-Meier Method
Description: rwPFS was defined as time (in months) from index date to death or disease progression (growth or worsening in the disease concluded by the treating clinician based on radiology, laboratory evidence, pathology, or clinical assessment) or end of record or end of data availability, whichever occurred first. If participants did not die or had disease progression, they were censored at the date of initiation of next line of therapy for participants with two or more lines of therapy or their last visit date for participants with only one line of therapy. Index date was defined as the start date of the first line therapy for Palbociclib + AI. Kaplan-Meier method was used for analysis.
Time Frame: From index date to death or disease progression or end of record/data availability or censored date, whichever occurred first, maximum up to approximately 43 months (data was retrieved and observed during 9 months of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + AI
Number analyzed (Participants) | 813
Months | 20.0 [17.3 to 22.2]

2. Secondary Outcome: Overall Survival (OS): Using Kaplan-Meier Method
Description: OS was defined as time (in months) from index date to the date of death. Participants who did not die during the period were censored at the time of data cut-off. Index date was defined as the start date of the first line therapy for Palbociclib + AI. Kaplan-Meier method was used for analysis.
Time Frame: From index date to death, maximum up to approximately 43 months (data was retrieved and observed during 9 months of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + AI
Number analyzed (Participants) | 813
Months | NA [NA to NA] — Median and 95% CI could not be estimated as there were less number of participants with the event.

3. Secondary Outcome: Number of Participants With Real World Tumour Response (rwTR)
Description: rwTR was determined based on complete response (CR), partial response (PR), stable disease (SD), progressive disease(PD), indeterminate and not documented. CR was defined as complete resolution of all visible disease. PR was defined as partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease. SD was defined as no change in overall size of visible disease; also included cases where some lesions increased in size and some lesions decreased in size. PD was determined based on growth or worsening in the disease concluded by the treating clinician based on radiology, laboratory evidence, pathology, or clinical assessment. Index date was defined as the start date of the first line therapy for Palbociclib + AI.
Time Frame: From index date to CR/PR/PD/SD pr PD, maximum up to approximately 43 months (data was retrieved and observed during 9 months of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + AI
Number analyzed (Participants) | 813
Participants
  CR | 67
  PR | 355
  SD | 166
  PD | 98
  Indeterminate | 17
  Not documented | 110

4. Secondary Outcome: Response Rate
Description: Response rate was defined as number of participants with complete response or partial response divided by the number of participants with at least one tumor assessment while on the index treatment. Index date was defined as the start date of the first line therapy for Palbociclib + AI. The result of this outcome measure was measured in terms of proportion of participants.
Time Frame: From index date to CR or PR, maximum up to approximately 43 months (data was retrieved and observed during 9 months of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Proportion of participants
Arm/Group | Palbociclib + AI
Number analyzed (Participants) | 813
Proportion of participants | 0.519

5. Secondary Outcome: Real-World Duration of Treatment (rwDOT): Using Kaplan-Meier Method
Description: rwDOT was defined as time (in months) from index treatment initiation to end of the treatment. Index date was defined as the start date of the first line therapy for Palbociclib + AI. Kaplan-Meier method was used for analysis.
Time Frame: From index treatment initiation up to end of treatment, maximum up to approximately 43 months (data was retrieved and observed during 9 months of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + AI
Number analyzed (Participants) | 813
Months | 16.3 [14.4 to 20.5]

6. Secondary Outcome: Time From Index Date to Next Line of Anti-Cancer Therapy: Using Kaplan-Meier Method
Description: The time (in months) from index treatment initiation to next line of anti-cancer therapy or death from any cause, whichever occurred first was reported in this outcome measure. Index date was defined as the start date of the first line therapy for Palbociclib + AI. Kaplan-Meier method was used for analysis.
Time Frame: From index treatment initiation up to next line of anti-cancer therapy or death from any cause, whichever occurred first, maximum up to approximately 43 months (data was retrieved and observed during 9 months of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + AI
Number analyzed (Participants) | 813
Months | 24.6 [22.0 to 26.4]

7. Secondary Outcome: Time to First Use of Chemotherapy: Using Kaplan-Meier Method
Description: The time (in months) from index treatment initiation to first use of chemotherapy or death from any cause, whichever occurred first was reported in this outcome measure. Index date was defined as the start date of the first line therapy for Palbociclib + AI. Kaplan-Meier method was used for analysis.
Time Frame: From index treatment initiation to first use of chemotherapy or death from any cause, whichever occurred first, maximum up to approximately 43 months (data was retrieved and observed during 9 months of this retrospective study)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib + AI
Number analyzed (Participants) | 813
Months | 36.6 [32.8 to NA] — Upper limit of 95% CI could not be reached due to less number of participants with event.

ADVERSE EVENTS:
Time Frame: All-cause mortality: from index date to death or disease progression or end of record/data availability or censored date, whichever occurred first, maximum up to approximately 43 months (data was retrieved and observed during 9 months of this retrospective study); Data for non-serious adverse events and serious adverse events (SAEs) were not collected and evaluated during the study; hence timeframe is not applicable for non-SAEs and SAEs
Description: Due to non-interventional nature of the study, data for non-SAEs and SAEs were not collected.
Arm/Group | Palbociclib + AI
All-Cause Mortality (participants affected / at risk) | 176/813
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-11-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT04176354/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT04176354/SAP_001.pdf